CLINICAL TRIAL: NCT06293781
Title: The Efficacy and Treatment Mechanisms of the Web-based Acceptance and Commitment Therapy for Patients with Major Depressive Disorder
Brief Title: Application of the Web-based Acceptance and Commitment Therapy for Depression
Acronym: ACTION
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gachon University (Other)
Responsible Party: Principal Investigator, Kyoung-Sae Na, Associate Professor, Gachon University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GachonU
Record Dates: First submitted 2024-02-18; First posted 2024-03-05 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-02

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ACT (Experimental): Web-based ACT with treatment as usual
  Interventions: Device: Web-based ACT; Behavioral: Treatment as usual
- Controls (Active Comparator): Waitlist being on the treatment as usual
  Interventions: Behavioral: Treatment as usual

INTERVENTIONS:
Device: Web-based ACT — ACT program delivered online
  Arms: ACT
Behavioral: Treatment as usual — Treatment as usual for major depressive disorder

SUMMARY:
PROSPECTIVE INTERVENTION STUDY; EFFICACY OF WEB-BASED ACCEPTANCE AND COMMITMENT THERAPY

DETAILED DESCRIPTION:
Acceptance Commitment Therapy (ACT) is known to help people recover from depression by improving psychological flexibility through acceptance, defusion, self-as-context, present moment, committed action, and helping them live a values-based life. This study is a randomized controlled trial to determine if web-based ACT leads to changes in the psychological flexibility and cognitive fusion. Also, through the functional MRI study, possible treatment mechanisms by which the web-based ACT exerts will be identified.

ELIGIBILITY:
Inclusion Criteria:

* Patients who diagnosed major depressive disorder

Exclusion Criteria:

* Patients who have serious medical problems, metal implants in their bodies, severe brain injury or brain disease
* Women who were pregnant or nursing
* Patients at high risk for suicide

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-12-19 (Actual); Primary Completion 2025-02-28 (Estimated); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
Acceptance and Action Questionnaire-II | 6 weeks
  Psychological flexibility
Hamilton Rating Scale for Depression | 6 weeks
  Interviewer-rated depression scale

SECONDARY OUTCOMES:
Cognitive Fusion Questionnaire | 6 weeks
  Cognitive fusion
Functional Connectivity | 6 weeks
  functional connectivity of the brain during resting state
Valuing | 6 weeks
  Measuring one's valuing
Beck Depression Inventory | 6 weeks
  Measuring subjective depression
Beck Anxiety Inventory | 6 weeks
  Measuring subjective anxiety
Beck Hopelessness Scale | 6 weeks
  Measuring hopelessness by the Beck Hopelessness Scale
Beck Scale for Suicide Ideation | 6 weeks
  Measuring suicidality

CONTACTS AND LOCATIONS:
Locations (1):
- Kyoung-Sae Na, Incheon, Please Incheon, South Korea

IPD SHARING:
Plan to Share IPD: No